CLINICAL TRIAL: NCT05055154
Title: Oxidative Stress and L-CBMN Cytome Assay Parameters Levels in Severely Obese With BMI ≥ 35kg/m2 After 3 Weeks 567 kcal Hospital Controlled VLCD
Brief Title: Oxidative Stress and L-CBMN Cytome Assay in Obese After 3 Weeks VLCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Special Hospital for Extended Treatment of Duga Resa (Other Government)
Collaborators: Institute for Medical Research and Occupational Health (Unknown); University of Zagreb (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSMN35aVLCD-26
Record Dates: First submitted 2021-09-14; First posted 2021-09-24 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Obesity; Weight Loss; DNA Damage
Keywords: Obesity; Very low calorie diet; Oxidative stress; Micronuclei; apoptosis
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Very low calorie diet (Experimental): Use of very low calorie diet prepared in the hospital
  Interventions: Device: Very low calorie diet

INTERVENTIONS:
Device: Very low calorie diet — In hospital patients will eat prepared diet with 567 kcal a day during 3 weeks

SUMMARY:
Obesity leads to physiological imbalance resulting in hyperglycemia, dyslipidaemia and inflammation and can generate systematic oxidative stress through multiple biochemical mechanisms. Oxidative stress (OS) can induce DNA damage and inhibit DNA repair mechanisms. Very low calorie diet (VLCD) have rapid positive effect on weight loss, glucose homeostasis, insulin resistance, inflammation and OS. The aim of this study is to determine the effect of a three-week VLCD on anthropometric, biochemical and genomic parameters in individuals with BMI ≥ 35kg/m2.

DETAILED DESCRIPTION:
Obesity is a complex chronic multifactorial disease associated with concomitant or increased risk for chronic inflammation, insulin resistance, dyslipidemia, oxidative stress, type 2 diabetes, cardiovascular disease, stroke and multiple cancer types. Oxidative stress (OS) can cause permanent DNA damage which could be detected with lymphocytes cytokinesis-block micronucleus (L-CBMN) cytome assay. Weight loss and improvement of dietary habits in people with obesity can affect genome stability and have beneficial effects on insulin sensitivity, inflammation and OS. Effects of very low calorie diet (VLCD) on DNA damage are scarce. The aim of this study is to determine the effect of a three-week VLCD used in Special Hospital for extended treatment of Duga Resa in patients with BMI ≥ 35kg/m2 on permanent DNA damage, lipid profile, insulin resistance, inflammation and anthropometric parameters.

ELIGIBILITY:
Inclusion Criteria:

* body mass index ≥ 35 kg/m2

Exclusion Criteria:

* pregnancy
* actual tumor diseases
* recent diagnostic or treatment exposures to ionizing radiation in the period of one year
* individuals not willing to stay 3 weeks under supervision under full 24 h surveillance from the medical stuff

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-06-14 (Actual); Primary Completion 2020-11-03 (Actual); Study Completion 2020-11-03 (Actual)

PRIMARY OUTCOMES:
The changes in body mass index | Baseline, after 3 weeks of VLCD
  Body mass index is calculated by dividing body mass (kg) with square of body height (m)
The changes in the body fat mass | Baseline, after 3 weeks of VLCD
  Body fat mass (kg) assessed with bioelectrical impedance method
The changes in the skeletal muscle mass | Baseline, after 3 weeks of VLCD
  Skeletal muscle mass (kg) assessed with bioelectrical impedance method
The changes in the percent body fat | Baseline, after 3 weeks of VLCD
  Percent body fat (%) assessed with bioelectrical impedance method
The changes in fasting glucose concentration | Baseline, after 3 weeks of VLCD
  Concentration of glucose (mmol/L)
The changes in urea concentration | Baseline, after 3 weeks of VLCD
  Concentration of urea (mmol/L)
The changes in lipid profile | Baseline, after 3 weeks of VLCD
  Concentrations of triglycerides (mmo/L), LDL (mmol/L), HDL (mmol/L) cholesterol (mmol/L)
The changes in insulin concentration | Baseline, after 3 weeks of VLCD
  Concentration of insulin (mIU/L)
The changes in homeostatic model assessment (HOMA) index | Baseline, after 3 weeks of VLCD
  HOMA index is calculated according to the following formula: glucose (mmol/L) x insulin (mIU/L)/22.5
The changes in inflammation parameters | Baseline, after 3 weeks of VLCD
  Concentration of C-reactive protein (mg/L) and total white blood cell count

SECONDARY OUTCOMES:
The changes in oxidative stress | Baseline, after 3 weeks of VLCD
  Concentration of glutathione (RFU) and reactive oxygen species (RFU)
The changes in DNA damage | Baseline, after 3 weeks of VLCD
  Frequency of micronucleus, nuclear buds, nucleoplasmic bridges, apoptotic and necrotic cells among 1000 lymphocytes

CONTACTS AND LOCATIONS:
Overall Officials: Mirta Milic, PhD, Principal Investigator — Institute for Medical Research and Occupational Health; Dragan Bozcevic, Doctor, Principal Investigator — Special Hospital for Extended Treatment of Duga Resa; Ana-Marija Domijan, Prof., Principal Investigator — University of Zagreb
Locations (1):
- Special Hospital for Extended Treatment of Duga Resa, Duga Resa, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grindel A, Brath H, Nersesyan A, Knasmueller S, Wagner KH. Association of Genomic Instability with HbA1c levels and Medication in Diabetic Patients. Sci Rep. 2017 Feb 2;7:41985. doi: 10.1038/srep41985. PMID 28150817
- [Background] Franzke B, Schwingshackl L, Wagner KH. Chromosomal damage measured by the cytokinesis block micronucleus cytome assay in diabetes and obesity - A systematic review and meta-analysis. Mutat Res Rev Mutat Res. 2020 Oct-Dec;786:108343. doi: 10.1016/j.mrrev.2020.108343. Epub 2020 Nov 2. PMID 33339574
- [Background] Mulligan AA, Luben RN, Bhaniani A, Parry-Smith DJ, O'Connor L, Khawaja AP, Forouhi NG, Khaw KT; EPIC-Norfolk FFQ Study. A new tool for converting food frequency questionnaire data into nutrient and food group values: FETA research methods and availability. BMJ Open. 2014 Mar 27;4(3):e004503. doi: 10.1136/bmjopen-2013-004503. PMID 24674997
- [Background] Kamencic H, Lyon A, Paterson PG, Juurlink BH. Monochlorobimane fluorometric method to measure tissue glutathione. Anal Biochem. 2000 Nov 1;286(1):35-7. doi: 10.1006/abio.2000.4765. PMID 11038270
- [Background] Kalyanaraman B, Darley-Usmar V, Davies KJ, Dennery PA, Forman HJ, Grisham MB, Mann GE, Moore K, Roberts LJ 2nd, Ischiropoulos H. Measuring reactive oxygen and nitrogen species with fluorescent probes: challenges and limitations. Free Radic Biol Med. 2012 Jan 1;52(1):1-6. doi: 10.1016/j.freeradbiomed.2011.09.030. Epub 2011 Oct 2. PMID 22027063
- [Background] Ustundag B, Gungor S, Aygun AD, Turgut M, Yilmaz E. Oxidative status and serum leptin levels in obese prepubertal children. Cell Biochem Funct. 2007 Sep-Oct;25(5):479-83. doi: 10.1002/cbf.1334. PMID 16874844
- [Background] Furukawa S, Fujita T, Shimabukuro M, Iwaki M, Yamada Y, Nakajima Y, Nakayama O, Makishima M, Matsuda M, Shimomura I. Increased oxidative stress in obesity and its impact on metabolic syndrome. J Clin Invest. 2004 Dec;114(12):1752-61. doi: 10.1172/JCI21625. PMID 15599400
- [Background] Keaney JF Jr, Larson MG, Vasan RS, Wilson PW, Lipinska I, Corey D, Massaro JM, Sutherland P, Vita JA, Benjamin EJ; Framingham Study. Obesity and systemic oxidative stress: clinical correlates of oxidative stress in the Framingham Study. Arterioscler Thromb Vasc Biol. 2003 Mar 1;23(3):434-9. doi: 10.1161/01.ATV.0000058402.34138.11. Epub 2003 Jan 30. PMID 12615693
- [Background] Il'yasova D, Wang F, Spasojevic I, Base K, D'Agostino RB Jr, Wagenknecht LE. Racial differences in urinary F2-isoprostane levels and the cross-sectional association with BMI. Obesity (Silver Spring). 2012 Oct;20(10):2147-50. doi: 10.1038/oby.2012.170. Epub 2012 Jun 22. PMID 22836686
- [Background] Kobayashi H, Matsuda M, Fukuhara A, Komuro R, Shimomura I. Dysregulated glutathione metabolism links to impaired insulin action in adipocytes. Am J Physiol Endocrinol Metab. 2009 Jun;296(6):E1326-34. doi: 10.1152/ajpendo.90921.2008. Epub 2009 Apr 14. PMID 19366877
- [Background] Tormos KV, Anso E, Hamanaka RB, Eisenbart J, Joseph J, Kalyanaraman B, Chandel NS. Mitochondrial complex III ROS regulate adipocyte differentiation. Cell Metab. 2011 Oct 5;14(4):537-44. doi: 10.1016/j.cmet.2011.08.007. PMID 21982713
- [Background] Won HY, Sohn JH, Min HJ, Lee K, Woo HA, Ho YS, Park JW, Rhee SG, Hwang ES. Glutathione peroxidase 1 deficiency attenuates allergen-induced airway inflammation by suppressing Th2 and Th17 cell development. Antioxid Redox Signal. 2010 Sep 1;13(5):575-87. doi: 10.1089/ars.2009.2989. PMID 20367278
- [Background] Bozinovski S, Seow HJ, Crack PJ, Anderson GP, Vlahos R. Glutathione peroxidase-1 primes pro-inflammatory cytokine production after LPS challenge in vivo. PLoS One. 2012;7(3):e33172. doi: 10.1371/journal.pone.0033172. Epub 2012 Mar 6. PMID 22412999
- [Background] Picklo MJ, Long EK, Vomhof-DeKrey EE. Glutathionyl systems and metabolic dysfunction in obesity. Nutr Rev. 2015 Dec;73(12):858-68. doi: 10.1093/nutrit/nuv042. Epub 2015 Oct 22. PMID 26493322
- [Background] Setayesh T, Misik M, Langie SAS, Godschalk R, Waldherr M, Bauer T, Leitner S, Bichler C, Prager G, Krupitza G, Haslberger A, Knasmuller S. Impact of Weight Loss Strategies on Obesity-Induced DNA Damage. Mol Nutr Food Res. 2019 Sep;63(17):e1900045. doi: 10.1002/mnfr.201900045. Epub 2019 Jun 14. PMID 31141317
- [Background] Santovito A, Gendusa C. Micronuclei frequency in peripheral blood lymphocytes of healthy subjects living in turin (North-Italy): contribution of body mass index, age and sex. Ann Hum Biol. 2020 Feb;47(1):48-54. doi: 10.1080/03014460.2020.1714728. Epub 2020 Jan 23. PMID 31969023
- [Background] Donmez-Altuntas H, Sahin F, Bayram F, Bitgen N, Mert M, Guclu K, Hamurcu Z, Aribas S, Gundogan K, Diri H. Evaluation of chromosomal damage, cytostasis, cytotoxicity, oxidative DNA damage and their association with body-mass index in obese subjects. Mutat Res Genet Toxicol Environ Mutagen. 2014 Sep 1;771:30-6. doi: 10.1016/j.mrgentox.2014.06.006. Epub 2014 Jun 28. PMID 25308439